CLINICAL TRIAL: NCT02514915
Title: Phase II Study Determining the Efficacy of Pre-operative Stereotactic Radiosurgery Followed by Resection for Brain Metastases
Brief Title: Pre-operative Stereotactic Radiosurgery Followed by Resection for Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Wilke (Other)
Responsible Party: Sponsor-Investigator, Christopher Wilke, Clinical Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 14-150
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Malignant Neoplasm Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Stereotactic Radiosurgery (Other): Subjects will receive stereotactic radiosurgery prior to resection
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Radiation therapy

SUMMARY:
The primary goal of this research study is to determine the efficacy of giving pre-operative radiosurgery to patients pending resection of a brain metastasis.

DETAILED DESCRIPTION:
Patients who have a brain metastasis surgically resected have very high local rates of disease relapse, and so the standard of care is to give either whole brain irradiation or stereotactic radiosurgery to the resection cavity in order to prevent disease recurrence. Stereotactic radiosurgery generally offers a more favorable side effect profile than whole brain irradiation, but targeting a surgical resection bed can be a challenge, as post surgical changes make it more difficult to distinguish residual tumor from scar, and much of the dose ends up being focused on the center of the resection cavity, where there are no substantial tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Karnofsky performance status of at least 50
* No contraindications to MRI scanning with intravenous contrast.
* MRI scan consistent with brain metastasis as per radiology report.
* Target lesion must measure at least 15 mm in at least one dimension, and no more than 4 cm in any dimension.
* Patients must have an extra-cranial primary tumor diagnosis.
* Patients will have no more than 4 distinct lesions within the brain. At least 1 lesion has been recommended for surgical removal based on size, symptomology, or regional mass effect on the brain.
* Additional lesions will each be treated with stereotactic radiosurgery.
* Patients with a documented symptomatic lesion size smaller than 3cm requiring clinical surgical resection
* Must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks and discomforts

Exclusion Criteria:

* Primary tumor histology of lymphoma, leukemia, multiple myeloma or germ cell tumor. Moribund status or status epilepticus.
* Supratentorial mass effect with greater than 5 mm of midline shift or hydrocephalus. Infratentorial mass effect with fourth ventricle effacement or hydrocephalus.
* More than four additional diagnosed brain metastases.
* Contraindication to general anesthesia.
* Adjacent tumor location to optic apparatus or brainstem, precluding achievement of meaningful dose with SRS.
* Primary brain tumor.
* Contraindication to MRI scans or intravenous contrast.
* Pregnant and breast-feeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Wilke, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Radiation Oncology Department, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.33333 (8.6359)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Local Control Rate (LCR) at 6 Months
Description: The probability that patients experience a change in size of a tumor (measured by the amount of space taken up by the tumor). Tumor volume was measured at 6 months compared to the tumor volume at the start of radiotherapy.
Time Frame: At 6 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 16
proportion of patients | 0.817 [0.669 to 0.997]

2. Primary Outcome: Local Control Rate (LCR) at 12 Months
Description: The probability that patients experience a change in size of a tumor (measured by the amount of space taken up by the tumor). Tumor volume was measured at 12 months compared to the tumor volume at the start of radiotherapy.
Time Frame: At 12 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
proportion of patients | 0.817 [0.669 to 0.997]

3. Primary Outcome: Local Control Rate (LCR) at 24 Months
Description: The probability that patients experience a change in size of a tumor (measured by the amount of space taken up by the tumor). Tumor volume was measured at 24 months compared to the tumor volume at the start of radiotherapy.
Time Frame: At 24 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
proportion of patients | 0.749 [0.579 to 0.973]

4. Secondary Outcome: 6-month Overall Survival (OS)
Description: The probability of patients being alive at 6 months after the beginning of treatment.
Time Frame: At 6 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 17
proportion of patients | 0.708 [0.548 to 0.916]

5. Secondary Outcome: 12-month Overall Survival (OS)
Description: The probability of patients being alive at 12 months after the beginning of treatment.
Time Frame: At 12 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
proportion of patients | 0.625 [0.458 to 0.852]

6. Secondary Outcome: 24-month Overall Survival (OS)
Description: The probability of patients being alive at 24 months after the beginning of treatment.
Time Frame: At 24 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
proportion of patients | 0.500 [0.335 to 0.746]

7. Secondary Outcome: Distant Intracranial Failure
Description: The probability of new brain metastases at 6 months identified via magnetic resonance imaging.
Time Frame: At 6 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
proportion of patients | 0.689 [0.521 to 0.912]

8. Secondary Outcome: Distant Intracranial Failure
Description: The probability of new brain metastases at 12 months identified via magnetic resonance imaging.
Time Frame: At 12 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 11
proportion of patients | 0.632 [0.455 to 0.877]

9. Secondary Outcome: Distant Intracranial Failure
Description: The probability of new brain metastases at 24 months identified via magnetic resonance imaging.
Time Frame: At 24 months
Population: All patients who received radiotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 8
proportion of patients | 0.502 [0.317 to 0.796]

10. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT - BR (FACT - BRAIN)
Description: The Functional Assessment of Cancer Therapy - Brain (FACT-Br) (23 questions that assess brain-tumor related issues) including the FACT-General (FACT-G), a core questionnaire used to determine the more general domains of QOL among all cancer patients was administered. This assessment is a 50 item, self-administered questionnaire used to assess Quality of Life, including, Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Subscale scores range from 0-4. FACT-G = (PWB - 7 items, score range 0-28) + (SWB - 7 items, score range 0-28) + (EWB - 6 items, score 0-24) + (FWB - 7 items, 0-28). The assessment takes 10-15 minutes to completed and is scored using a 5-point Likert-type scale. FACT Gen Scores range from 0-108. Brain (FACT-Br) Scores range from 0-92 (23 questions with 0-4 score). Thus, total assessments combine scores range from 0-200. Higher total scores indicating better quality of life.
Time Frame: At 6 months (1.5-month window)
Population: All patients who received radiotherapy and completed required surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 5
score on a scale | 139.878 (20.59528024)

11. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT - BR (FACT - BRAIN)
Description: as for outcome 10
Time Frame: At 6 months (3-month window)
Population: All patients who received radiotherapy and completed required surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 11
score on a scale | 142.1581538 (23.8429411)

12. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT - BR (FACT - BRAIN)
Description: as for outcome 10
Time Frame: At 12 months (1.5-month window)
Population: All patients who received radiotherapy and completed required surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 6
score on a scale | 141.0952857 (26.95376082)

13. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT - BR (FACT - BRAIN)
Description: as for outcome 10
Time Frame: At 12 months (3-month window)
Population: All patients who received radiotherapy and completed required surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 7
score on a scale | 143.3974615 (23.28519091)

14. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT - BR (FACT - BRAIN)
Description: as for outcome 10
Time Frame: At 24 months (1.5-month window)
Population: All patients who received radiotherapy and completed required surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 1
score on a scale | 167 (NA) — Single participant score; no SD

15. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT - BR (FACT - BRAIN)
Description: as for outcome 10
Time Frame: At 24 months (3-month window)
Population: All patients who received radiotherapy and completed required surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 5
score on a scale | 150.1484545 (23.94648714)

ADVERSE EVENTS:
Time Frame: Patients were monitored for Adverse Events for up to 60 days post treatment. Adverse events data were collected for 2 years, 10 months. Deaths were assessed for up to 55 months.
Arm/Group | Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 19/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT02514915/Prot_SAP_000.pdf